CLINICAL TRIAL: NCT03836326
Title: Developmental Outcome of Preterm Infants Enrolled in a Randomized Clinical of a Parent Administered Sensorimotor Intervention in the Neonatal Intensive Care Unit
Brief Title: A Parent Administered Sensorimotor Intervention and Developmental Outcome of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sandra Fucile (Other)
Responsible Party: Sponsor-Investigator, Dr. Sandra Fucile, PI, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 6023834
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Premature Infant; Developmental Delay
Keywords: Prematurity; Development; Parental engagement; Parental satisfaction
MeSH Terms: conditions — Premature Birth; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Randomized clinical trail
Masking Description: A prospective randomized block clinical trial will be conducted. Infants will be randomized into experimental (PASI program) and control (standard care program) groups using a block size of four per arm, where the first set of four participants will be in the experimental group and once they have completed the intervention, the subsequent set of four participants will be in the control group. A randomized block design was selected because the treatment assignment cannot be masked. The block randomization procedure will reduce the potential for contamination between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor intervention (Experimental): Is a 15-minute intervention consisting of tactile (i.e., stroking the whole body) and oral input (i.e., stroking the oral structures) for 15 minutes duration. The program will start 24 hours after nasal continuous positive airway pressure (NCPAP) is discontinued and 24 hours after 80 ml/kg/day of enteral feeds are tolerated. The program will be administered once a day for 10 days, within a 14-day period. The parents will perform all the interventions in the NICU. The infants will remain in the isolette for the duration of the program. This intervention does not involve any drugs or medical procedures. It is an intervention commonly used by occupational and physical therapists in the neonatal intensive care unit.
  Interventions: Other: Sensorimotor intervention; Other: Story telling attention refocusing intervention
- Control (Other): Infants in the control group will receive standard care only.
  Interventions: Other: Control

INTERVENTIONS:
Other: Sensorimotor intervention — Sensorimotor intervention involves, stroking of the whole body including the oral structures, trunk and limbs. This intervention does not involve any drugs or medical procedure.
  Other Names: Supplemental stimulation; Sensory input; Tactile input; Oral input
  Arms: Sensorimotor intervention
Other: Control — Routine care provided by health professionals in the NICU
  Arms: Control
Other: Story telling attention refocusing intervention — A contact-free intervention where parents share stories with their infant for 10 minutes 3 times per week.
  Other Names: STAR
  Arms: Sensorimotor intervention

SUMMARY:
Advances in medical technologies over the last three decades have increased survival rates in infants born preterm . Preterm infants are at high risk of developing developmental delays. Implementation of effective strategies aimed at improving the developmental outcome of preterm born children is critical.

The proposed study is designed to evaluate the addition of a parent administered sensorimotor program on the developmental outcome of infants who are born preterm.

DETAILED DESCRIPTION:
Children who are born prematurely are at a higher risk of developing developmental delays than children born at term. Early experiences in the neonatal intensive care unit (NICU) can influence developmental outcomes. Sensorimotor interventions as well as parental engagement have been designed with the aim of improving the development of children born preterm. Substantial evidence supports the benefits of each intervention on improving developmental outcomes. However, there remains a significant gap in the literature on the efficacy of a parent administered sensorimotor intervention (PASI) program in the NICU on infant's development. The proposed study is designed to evaluate the potential benefits of such a program on infant's development. A randomized block clinical trial will be performed.

A total of 84 preterm infants (< 34 weeks gestation) will be recruited and randomized. Infants in the experimental group will receive the sensorimotor program,consisting of tactile (whole body) and oral input for 15 minutes, one time per day, for 10 days. Infants in the control group will receive standard care. The following outcomes will be monitored time to attainment of complete oral feeds (primary outcome), rate of weight gain, length of hospitalization, and developmental outcomes at 36 weeks corrected gestational age and at 4, 8, 12, 18 and 24 months corrected age. Results from this study will provide us with further knowledge on the impact of sensorimotor intervention on infants' developmental outcome as well as the effect of active parental involvement on infants' development. Provision of a PASI program is a safe and low cost effective intervention that may increase the development and quality of life of preterm born children and their family.

ELIGIBILITY:
Inclusion Criteria:

* Infants born < 34 weeks gestation
* Infants whose parent (s) intend on visiting regularly (> 5 days)

Exclusion Criteria:

* Infants born with a metabolic disorder or congenital abnormality
* Infants whose parents are unable to participate due to cognitive, physical or social issues.

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Attainment of independent oral feeds | 3 years
  Number of days to transition from complete tube to complete oral feeds.

SECONDARY OUTCOMES:
Weight gain | 3 years
  Weight gain velocity from start of study until hospital discharge
Length of hospital stay | 3 years
  Number of days from birth to discharge home
Test of infant motor performance | 3 years
  A standardized assessment measuring postural control and motor function in infants from 32 weeks gestation to 4 months corrected gestational age. Total raw scores range from 0-142, higher scores represent better motor function.
Acute stress of parents | 3 years
  The PSS: NICU assessment was used to assess acute stress of parents

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Fucile, PhD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No